CLINICAL TRIAL: NCT06982781
Title: A Retrospective Post-Market Clinical Study of the Flow Re-Direction Endoluminal Device System in the Treatment of Intracranial Aneurysms
Brief Title: FRED Retrospective Study of Intracranial Aneurysms Treatment
Acronym: FRED
Status: Not yet recruiting | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1106094
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Flow Re-Direction Endoluminal Device System(FRED) — Flow Diverter (FD) devices are developed based on reconstructing the parent artery's lumen. FDs are designed with a denser mesh compared to conventional intracranial stents. By covering the aneurysm neck, these stents redirect blood flow away from the aneurysm, promoting intra-aneurysmal flow stagnation and subsequent thrombosis formation. Currently, FDs are primarily used for the treatment of wide-neck aneurysms.

SUMMARY:
To evaluate the long-term safety and efficacy of Flow Re-Direction Endoluminal Device System (FRED) in the treatment of intracranial aneurysms in the post-market environment

DETAILED DESCRIPTION:
Study Objective: To evaluate the long-term safety and efficacy of Flow Re-Direction Endoluminal Device System (FRED) in the treatment of intracranial aneurysms in the post-market.

Study Design: Post-market, retrospective, multi-center, observational clinical study Study Population: Patient who has implanted at least one observational device in China mainland.

ELIGIBILITY:
Inclusion Criteria:

* People in China mainland who have been treated with FRED. The patients for whom clinical data are available

Exclusion Criteria:

* Patients who met the inclusion criteria at all time points were required to be included in the study. Therefore, no specific exclusion criteria were set.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has implanted at least one observational device in China mainland
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
O'Kelly-Marotta, OKM grade (Imaging Evaluation of a Target Aneurysm) | 6 month, 1 year
  Based on the evaluation of imaging results, the treatment of aneurysms was classified according to the following criteria. Digital Subtraction Angiography (DSA), Magnetic Resonance Angiography (MRA), or Computed Tomography Angiography (CTA) are acceptable, and it is recommended base CTA. The purpose of imaging follow-up information collection is to observe the effect of on the long-term closure of the aneurysm after treatment. Complete closure of the aneurysm would be associated with increased safety.
Raymond-Roy Grade (Adequate Occlusion Rate of Target Aneurysm) | 6 month, 1 year
  Adequate Occlusion is defined as Raymond-Roy Grade I or Grade II on imaging evaluation of the target aneurysm.
Technical Success rate | Immediate post-procedure
  The technical success rate refers to the proportion of technically successful patients in the total number of patients. Technical success is defined as successful stent placement and meet following criteria: Stent fully cover the aneurysm neck; Good wall apposition; Perfusion of the parent artery; Retention of contrast agent within the aneurysm;
Re-sheathing performance | Immediate post-procedure
  During procedure, the observational device can be retrieved / re-sheathed into the microcatheter and re-deployed at the desired target location or removed completely from the patient. But it must not be re-deployed more than three times. Re-sheath performance refers to the retrieving and re-deploying of observational device recorded during the procedure. Information such as the number of recoveries and the number of re-sheathings, the success rate of re-opening and other information are recorded to evaluate the re-sheath performance of the observational device.
Modified Rankin Scale (mRS) | 6 month, 1year
  The modified Rankin (mRS) score was used to evaluate the improvement of neurological function. The modified Rankin score assesses the ability to live independently in patients with Neurological disease [6]. There are 7 levels of this score, 0 points represent no symptoms of disability, higher scores mean worse prognosis of patients, and 6 points represent death, See the table below for detailed scores.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxiao Li, Principal Investigator — Henan Provincial People's Hospital; Sheng Guan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

DOCUMENTS (1):
  • Study Protocol (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT06982781/Prot_000.pdf